CLINICAL TRIAL: NCT01803711
Title: A Randomized, Double-Blind Placebo-controlled Study Evaluating the Efficacy of Omega 3 Fatty Acid Augmentation of Desvenlafaxine for the Treatment of Major Depressive Disorder in Patients With Medical Illness.
Brief Title: Omega 3 FA Supplements as Augmentation in the Treatment of Depression
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of recruitment and no resources
Sponsor: UConn Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OmegaDVS
Record Dates: First submitted 2013-02-28; First posted 2013-03-04 (Estimated); Results first posted 2017-12-27 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-11

CONDITIONS: Major Depression; Cancer; Diabetes; Cardiovascular Diseases
Keywords: Omega 3 fatty acid; Fish oil; Depression; cancer; diabetes; high blood pressure; cardiovascular
MeSH Terms: conditions — Depressive Disorder, Major; Neoplasms; Diabetes Mellitus; Cardiovascular Diseases; Depression; Hypertension | interventions — Desvenlafaxine Succinate; Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Desvenlafaxine + Omega 3 FA supplement (Experimental): Desvenlafaxine 50mg/day & Omega 3 FA supplement (range 2.4 gm/day - 4.8 gm day) over a 12 week period
  Interventions: Drug: Desvenlafaxine; Dietary Supplement: Omega 3 Fatty acids
- Desvenlafaxine + Placebo (for Omega 3 FA supplement) (Active Comparator): Desvenlafaxine 50mg/day & Placebo (for Omega 3 FA supplement) over a 12 week period
  Interventions: Drug: Desvenlafaxine; Drug: Placebo (for Omega 3 fatty acid supplement)

INTERVENTIONS:
Drug: Desvenlafaxine
  Other Names: Pristiq
Dietary Supplement: Omega 3 Fatty acids
  Arms: Desvenlafaxine + Omega 3 FA supplement
Drug: Placebo (for Omega 3 fatty acid supplement)
  Arms: Desvenlafaxine + Placebo (for Omega 3 FA supplement)

SUMMARY:
To assess the efficacy of Omega 3 Fatty acid (Omega 3 FA) augmentation of desvenlafaxine (DVS) compared to placebo augmentation of DVS when used to treat depression and anxiety symptoms in patients with select medical conditions (cancer, cardiovascular diseases and diabetes).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosed with depression and have cardiovascular disease, diabetes or cancer.
* Able to provide written informed consent prior to initiation of any study-related procedures.
* Able to understand and comply with the requirements of the study.

Exclusion Criteria:

* Hospitalized patients or psychotherapy for depression begun within 4 weeks.
* Patients with medically reversible causes of depression (e.g. hypothyroidism).
* Patients with significant comorbid symptoms (e.g. pain, insomnia) that have a direct causal relation to depressive and anxiety symptoms with these comorbid symptoms dominating the clinical scenario. Patients will be enrolled in the study if these comorbid symptoms merely coexist with depressive and anxiety symptoms and are not dominating the clinical scenario as judged by the study investigator
* Patients with an identifiable diagnosis of substance abuse or dependence within 6 months prior to evaluation (except those in full remission, or those with caffeine or nicotine dependence) as defined by DSM-IV criteria.
* Patients with any clinically significant unstable or inadequately treated co-morbid medical condition which, in the opinion of the investigator, would make the patient unsuited for the study
* Patients with currently active or with significant history of other clinically significant psychiatric disorders such as bipolar disorder, schizophrenia etc.
* Pregnant patients, breastfeeding or those planning to become pregnant during the study.
* Any other condition, which, in the opinion of the investigator, would make the patient, unsuited for enrollment in the study, including known or suspect history of allergy to fish oil, fish or desvenlafaxine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jayesh Kamath, MD PhD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 30 subjects underwent phone screening. Of these, a total of 6 subjects were consented and 5 met study eligibility criteria.
Pre-assignment Details: One subject who was consented did not meet the threshold for depression symptomatology during screening as determined by the Hospital Anxiety and Depression Scale.
Groups:
- Desvenlafaxine + Omega 3 FA Supplement: Desvenlafaxine 50mg/day & Omega 3 FA supplement (range 2.4 gm/day - 4.8 gm day) over a 12 week period
  Desvenlafaxine
  Omega 3 Fatty acids
  2 subjects were randomized to this group
- Desvenlafaxine + Placebo (for Omega 3 FA Supplement): Desvenlafaxine 50mg/day & Placebo (for Omega 3 FA supplement) over a 12 week period
  Desvenlafaxine
  Placebo (for Omega 3 fatty acid supplement)
  3 subjects were randomized to this group
Period: Overall Study
Arm/Group | Desvenlafaxine + Omega 3 FA Supplement | Desvenlafaxine + Placebo (for Omega 3 FA Supplement)
Started | 2 | 3
Completed | 1 | 2
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Desvenlafaxine + Omega 3 FA Supplement: Desvenlafaxine 50mg/day & Omega 3 FA supplement (range 2.4 gm/day - 4.8 gm day) over a 12 week period
  Desvenlafaxine
  Omega 3 Fatty acids
  Age range: 53 to 66 years Gender: 1 male and 1 female
- Desvenlafaxine + Placebo (for Omega 3 FA Supplement): Desvenlafaxine 50mg/day & Placebo (for Omega 3 FA supplement) over a 12 week period
  Desvenlafaxine
  Placebo (for Omega 3 fatty acid supplement) Age range: 53 to 66 years ] Gender: 1 male and 2 females
- Total: Total of all reporting groups
Arm/Group | Desvenlafaxine + Omega 3 FA Supplement | Desvenlafaxine + Placebo (for Omega 3 FA Supplement) | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 1 | 1 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  White Non-Hispanic/Latino | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Hospital Anxiety and Depression Scale
Description: Hospital Anxiety and Depression Scale: This is a validated scale for measuring depression/anxiety symptoms in patients with medical conditions.
Time Frame: 12 weeks from baseline
Population: Planned statistical analyses were not performed due to lack of adequate sample size. The data collected were not intended to be summarized if there were fewer than 10 participants.
Groups:
- Desvenlafaxine + Omega 3 FA Supplement: Desvenlafaxine 50mg/day & Omega 3 FA supplement (range 2.4 gm/day - 4.8 gm day) over a 12 week period
  Desvenlafaxine
  Omega 3 Fatty acids
- Desvenlafaxine + Placebo (for Omega 3 FA Supplement): Desvenlafaxine 50mg/day & Placebo (for Omega 3 FA supplement) over a 12 week period
  Desvenlafaxine
  Placebo (for Omega 3 fatty acid supplement)
Arm/Group | Desvenlafaxine + Omega 3 FA Supplement | Desvenlafaxine + Placebo (for Omega 3 FA Supplement)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Arm/Group | Desvenlafaxine + Omega 3 FA Supplement | Desvenlafaxine + Placebo (for Omega 3 FA Supplement)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Short Form Health Survey (SF-12)
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Arm/Group | Desvenlafaxine + Omega 3 FA Supplement | Desvenlafaxine + Placebo (for Omega 3 FA Supplement)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Visual Analog Scale for Energy (VAS-E)
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Arm/Group | Desvenlafaxine + Omega 3 FA Supplement | Desvenlafaxine + Placebo (for Omega 3 FA Supplement)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Visual Analog Scale for Pain (VAS-P)
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Arm/Group | Desvenlafaxine + Omega 3 FA Supplement | Desvenlafaxine + Placebo (for Omega 3 FA Supplement)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Leeds Sleep Evaluation Questionnaire (LSEQ)
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Arm/Group | Desvenlafaxine + Omega 3 FA Supplement | Desvenlafaxine + Placebo (for Omega 3 FA Supplement)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Desvenlafaxine + Omega 3 FA Supplement | Desvenlafaxine + Placebo (for Omega 3 FA Supplement)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 1/2 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desvenlafaxine + Omega 3 FA Supplement (N=2) | Desvenlafaxine + Placebo (for Omega 3 FA Supplement) (N=3)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Stomach upsets
Memory problems (Nervous system disorders) | 0 (0) | 1 (1) — Memory problems

LIMITATIONS AND CAVEATS:
Due to very low enrollment in both arms, only descriptive analyses was completed for both arms

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes